CLINICAL TRIAL: NCT01896271
Title: A Phase II Trial of High Dose IL-2 and Stereotactic Ablative Body Radiation Therapy (SABR) for Patients With Metastatic Clear Cell Renal Cell Cancer (mRCC)
Brief Title: High Dose IL-2 and Stereotactic Ablative Body Radiation Therapy for Metastatic Renal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Prometheus Laboratories (Industry)
Responsible Party: Principal Investigator, Raquibul Hannan, Principal Investigator, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 012013-041
Record Dates: First submitted 2013-07-05; First posted 2013-07-11 (Estimated); Results first posted 2021-08-23 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-07

CONDITIONS: Metastatic Clear Cell Renal Cell Carcinoma
Keywords: kidney cancer; metastatic cancer
MeSH Terms: conditions — Clear-cell metastatic renal cell carcinoma; Kidney Neoplasms; Neoplasm Metastasis | interventions — Interleukin-2; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- treatment (Experimental): HD IL-2 (brand name Proleukin), 600,000 U/kg q8h X 14 dose, IV infusion; SABR dose varying from 8Gy-20Gy in 1-3 fractions.
  Interventions: Drug: IL-2; Radiation: Stereotactic Ablative Body Radiation Therapy

INTERVENTIONS:
Drug: IL-2 — HD IL-2 (brand name Proleukin), 600,000 U/kg q8h X 14 dose, IV infusion
Radiation: Stereotactic Ablative Body Radiation Therapy — SABR dose varying from 8Gy-20Gy in 1-3 fractions
  Other Names: SABR, SBRT

SUMMARY:
In this i-SABR (immunotherapy + Stereotactic Ablative Body Radiation) trial, the stereotactic radiation to multiple metastatic sites is delivered not only to eradicate sites of bulky progressive disease, but also to provide antigen presentation and immune stimulation which is expected to act synergistically when immediately followed by the non-specific immune stimulation provided by treatment with HD IL-2 and thereby increase the response rate and complete response for metastatic clear cell renal cell cancer patients. Both HD IL-2 and SABR are FDA approved therapeutic cancer treatment

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy-proven metastatic clear cell RCC.
2. Radiographic evidence of metastatic disease. 2.1 Patients with any number of metastatic site are allowed to enroll. However, only up to six sites will be selected for SBRT treatment, at the discretion of the treating radiation oncologist.
3. Patient must have ≥1 lesion of size >1.5cm.
4. Previous treatment with surgery, radiation, chemotherapy, immunotherapy or any targeted agents are allowed 28 days before the start of HD IL-2
5. Age ≥ 18 years.
6. Performance status ECOG 0, 1.
7. Patient must be eligible for HD IL-2 treatment
8. Patient must be eligible for SABR to one or more extra cranial sites.
9. Adequate organ and marrow function as defined below:

   * leukocytes ≥ 3,000/mcL
   * absolute neutrophil count ≥ 1,500/mcL
   * platelets ≥ 50,000/mcl
   * total bilirubin ≤ 2mg/dL
   * AST(SGOT)/ALT(SPGT) ≤ 2.5 X institutional upper limit of normal
10. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

    10.1 A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:
    * Has not undergone a hysterectomy or bilateral oophorectomy; or
    * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
11. Ability to understand and the willingness to sign a written informed consent
12. Adequate Renal function with Cr ≤ 1.6 mg/dL.
13. Adequate cardiac function (adequate perfusion; no ischemia) on thallium (or Tc) stress test
14. Adequate pulmonary function on PFT (FEV1 >65%; DLCO>60%).

Exclusion Criteria:

1. Subjects who have had chemotherapy or radiotherapy within 4 weeks prior to entering the study
2. History of HIV, Hepatitis B, Hepatitis C and HTLV serology
3. Subjects may not be receiving any other investigational or standard antineoplastic agents.
4. Subjects with known brain metastases should be excluded from this clinical trial because of their poor prognosis
5. Subjects with life expectancy < 6 months.
6. History of allergic reactions to recombinant IL-2
7. Uncontrolled recurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia,.
8. Psychiatric illness/social situations that would limit compliance with study requirements.
9. Subjects must not be pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants.
10. Systemic or topical steroid use or other immunosuppressive therapy within the past 28 days
11. Subjects required to take corticosteroids or other immunosuppressive therapy such as those with organ allograft

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-10-02 (Actual); Primary Completion 2020-08-25 (Actual); Study Completion 2021-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raquibul Hannan, MD, PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment
Started | 30
Completed | 20
Not Completed | 10
Not completed — Physician Decision | 10

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 30
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 51.5 [47 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 25
  Non-white | 5

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: Treatment response will be measured using the immune related Response Evaluation Criteria in Solid Tumors (RECIST) criteria (iRECIST) which are a minor modification of RECIST 1.1 for immunotherapy
Time Frame: 6 months
Population: There were 5 patients without measurable disease at baseline and 5 additional patients without 2nd scan to confirm progression. Hence, they were not analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 20
Participants | 4

2. Secondary Outcome: Overall Survival
Description: Overall Survival (OS), which is defined as the time between date of registration and the date of death due to any cause.
Time Frame: 4 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment
Number analyzed (Participants) | 30
months | 39 [16 to 53]

3. Secondary Outcome: Progression Free Survival
Description: Progression Free Survival (PFS), which is defined according to the immune Response Evaluation Criteria in Solid Tumors (iRECIST) as the time between date of registration and the first date of documented disease progression or date of death due to any cause.
Time Frame: 4 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment
Number analyzed (Participants) | 20
months | 2.5 [2 to 8]

4. Secondary Outcome: Time to Progression
Description: Time to Progression (TTP), which is defined as time between date of registration and date of documented progression
Time Frame: 4 years
Population: This outcome measure was inadvertently added at the time of registration. This is same as progression free survival and measures and reports the exact same thing and is redundant. No separate data was collected from participants for this specific measure.
Arm/Group | Treatment
Number analyzed (Participants) | 0

5. Secondary Outcome: Local Control Rate
Description: Local recurrence is defined as tumor recurrence within the planning target volume. Local control rate will be evaluated by imaging techniques such as CT or MRI. Local recurrence will be defined as an increase of > 20% in tumor size.
Time Frame: 4 years
Measure: Number; unit: lesions
Units Other Than Participants: lesions
Arm/Group | Treatment
Number analyzed (Participants) | 30
Number analyzed (lesions) | 31
lesions | 30

6. Secondary Outcome: Median Response Duration
Description: Median response duration, which is defined as the time between the date a response (CR or PR) was first seen until date of progression
Time Frame: 4 years
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Treatment
Number analyzed (Participants) | 20
months | 26.7 [11.4 to 36.4]

7. Secondary Outcome: Tumor-specific Immune Response
Description: Immune response will be measured using ELISpot assay, T-cell proliferation assay and ELISA.
Time Frame: 4 years
Population: This data were never collected from the participants.
Arm/Group | Treatment
Number analyzed (Participants) | 0

8. Secondary Outcome: Number of Participants With Adverse Events
Description: Adverse events will be determined according to Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0.
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 30
Participants | 30

9. Secondary Outcome: Health-related Quality of Life (HRQoL).
Time Frame: 4 years
Population: The data were never collected from the participants.
Arm/Group | Treatment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 4 years
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 19/30
Serious Adverse Events (participants affected / at risk) | 22/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=30)
Cardiac (Cardiac disorders) | 3
Gastrointestinal (Gastrointestinal disorders) | 1
Hematology Coagulation (Blood and lymphatic system disorders) | 8
Hepatobiliary disorders (Hepatobiliary disorders) | 3
Hypotension (Cardiac disorders) | 2
Infection (Infections and infestations) | 3
Neurologic (Nervous system disorders) | 1
Other (General disorders) | 1
Renal/electrolytes (Renal and urinary disorders) | 11
Respiratory (Respiratory, thoracic and mediastinal disorders) | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=30)
Cardiac (Cardiac disorders) | 22
Constitutional (General disorders) | 27
Gastrointestinal (Gastrointestinal disorders) | 22
Hematology Coagulation (Blood and lymphatic system disorders) | 28
Hypotension (Cardiac disorders) | 18
Infection (Infections and infestations) | 5
Neurologic (Nervous system disorders) | 12
Other (General disorders) | 14
Psychiatric (Psychiatric disorders) | 6
Renal/electrolytes (Renal and urinary disorders) | 29
Respiratory (Respiratory, thoracic and mediastinal disorders) | 13
Skin (Skin and subcutaneous tissue disorders) | 21
Hepatobiliary disorders (Hepatobiliary disorders) | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-05-20): https://cdn.clinicaltrials.gov/large-docs/71/NCT01896271/Prot_SAP_000.pdf
  • Informed Consent Form (2019-05-20): https://cdn.clinicaltrials.gov/large-docs/71/NCT01896271/ICF_001.pdf